CLINICAL TRIAL: NCT03984552
Title: Validation of Rapid Tests for the Serological Diagnosis of HIV in 9 to 24 Months Old Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Other Study IDs: ASCLIN 002/2012
Record Dates: First submitted 2019-06-11; First posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Human Immunodeficiency Virus Transmission; Human Immunodeficiency Virus; Diagnoses, Syndromes, and Conditions
Keywords: HIV; rapid test; HIV infection; vertical transmission
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Disease; HIV Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — First, a sample of oral fluid for the RT DPP HIV 1/2 will be harvested.Then, the blood from the finger stick will be used to perform RT DPP HIV 1 / 2 ® and rapid imunoblot HIV 1/ 2(IB).The results of the rapid tests will be available in up to 30 minutes and will be recorded in specific forms for further analysis of concordance with the molecular results. The blood samples and parts of them (serum and plasma) collected in this study will be used only for the examinations foreseen in this research project and will be kept under the responsibility of the researcher Dr. Luiz Antonio Bastos Camacho in Bio-Manguinhos / Fundação Oswaldo Cruz for 10 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: This was an observational study of medical devices (rapid tests) used for the HIV diagnosis in children up to 2 years — These rapid tests are based on lateral flow immunochromatography technology, in which a nitrocellulose membrane is impregnated with the antigen of interest. The patient sample (blood, serum, plasma, oral fluid, etc.) is applied in this membrane which facilitates the interaction of antibodies in the sample with the antigens on the membrane. This reaction becomes visible to the naked eye thanks to a color developing revelator.
  The entire testing process, from sample collection to result reading takes no more than 40 minutes and does not depend on laboratory facilities.

SUMMARY:
Antiretroviral therapy of the mother and of the newborn associated with alternative schemes of breastfeeding can reduce these transmission rates to 1%. The diagnosis of HIV infection in newborns is based on PCR for detection of viral genetic material, a procedure that is expensive and of complex logistics. Tests based on detection of antibodies are faster and cheaper but cannot distinguish infected child or maternal antibodies passed to the fetus through the placenta. Nevertheless, the so-called rapid tests have been implemented in the network of health services because of their simplicity and performance comparable to conventional tests. DPP HIV 1/2 test, produced by Bio-Manguinos/Fiocruz, usage is limited by the manufacturer to over 24 months of age children, though the guidelines control programs already recommend the use from 18 months in Brazil and 9 months in other countries. Data on the accuracy of the rapid test under 24 months of age are scarce. This proposal aims to assess the performance of rapid tests produced by Bio-Manguinhos in diagnostic protocols for HIV infection in children 9-24 months old, in order to obtain empirical data to support the current recommendations on rapid tests, particularly in countries with limited access to tests that require specialized laboratories. The validation of rapid HIV testing in other age groups is a requirement of the national regulatory authorities, and has important implications for programs to control HIV-AIDS in populations from countries with limited access to specialized laboratory resources. The use of the rapid test can also represent a significant reduction in costs, as it allows limiting the use of molecular tests to complex and expensive confirmation cases.

DETAILED DESCRIPTION:
It concerns a study with a sample composed of children born from HIV positive mothers, age between 9 and 24 months old, with confirmed or discarded infection for HIV determined by molecular testing. Samples from the volunteers will be subjected to rapid tests and serological and molecular reference tests.

After obtaining consent from the child's guardian,a brief interview will take place with completing the questionnaire of inclusion in the research. Then, the collection of fluid in the oral cavity as well as the fingerstick puncture will be conducted for the HIV rapid tests procedures.

The results of the rapid tests will be compared with the ones from the molecular testing and the concordance will be determined for each age group separately.

The study has being conducted by four clinical research sites at Brazil, distributed in three different states, and a clinical research site at Tanzânia: Instituto Fernandes Figueira (IFF - Fiocruz) at Rio de Janeiro; Hospital Geral de Nova Iguaçu (HGNI) at Rio de Janeiro, Fundação de Medicina Tropical Doutor Heitor Vieira Dourado (FMT-HVD) at Amazonas; Secretaria de Estado de Saúde Pública do Pará (URES - Materno Infantil - UREMIA) at Pará and National Institute for Medical Research (NIMR) at Tanga in Tanzania.

ELIGIBILITY:
Inclusion Criteria:

Children must be born from a HIV infected mother; Molecular diagnostic tests available.

Exclusion Criteria:

Not applicable

Ages: 9 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 502 children born from a HIV infected mother, divided in the following groups:
  1. 251 HIV infected children, divided in the following subgroups:
     1. 9-15 months old;
     2. 16-21 months old;
     3. 22-24 months old
  2. 251 HIV non infected children, divided in the following subgroups:
     1. 9-15 months old;
     2. 16-21 months old;
     3. 22-24 months old
Sampling Method: Probability Sample
Enrollment: 502 (Estimated)
Dates: Start 2015-03-12 (Actual); Primary Completion 2020-06-05 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the Bio-Manguinhos / Fiocruz Rapid DPP® HIV-1/2 Immunoblot | Day 1
  Sensitivity and specificity of the Bio-Manguinhos / Fiocruz Rapid DPP® HIV-1/2 Immunoblot, based on the molecular test.

SECONDARY OUTCOMES:
Efficacy of the Bio-Manguinhos / Fiocruz HIV-1/2 rapid serum screening test | Day 1
  Sensitivity and specificity of the Bio-Manguinhos / Fiocruz HIV-1/2 rapid serum screening test in children aged 9 to 24 months, using the Elisa or chemiluminescence and molecular test as reference.
Efficacy of the rapid Oral Fluid test HIV- 1/2 Bio- Manguinhos | Day 1
  Sensitivity and specificity of the rapid Oral Fluid test HIV- 1/2 Bio- Manguinhos in children ,taking as reference molecular testing.
Variations in the accuracy of rapid tests | Day 1
  Covariables of mothers and children

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Antonio B Camacho, DrPH, Principal Investigator — Escola Nacional de Saúde Pública - ENSP/Fiocruz
Locations (1):
- Assessoria Clinica / Bio-Manguinhos / Fiocruz, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No